CLINICAL TRIAL: NCT02505880
Title: Evaluation of Perioperative Use of Hypnosis in Pediatric Surgery: Clinical and Medico-economic Interests
Brief Title: Hypnosis Versus General Anesthesia in Pediatric Surgery: Clinical and Medico-economic Interests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9518; 2014-A01776-41 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-06-15; First posted 2015-07-22 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2015-07

CONDITIONS: Minimally Invasive Surgery
Keywords: Hypnosis; Pediatric surgery; Anesthesia
MeSH Terms: interventions — Anesthetics, Local; Hypnosis; Anesthesia, General

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: General anesthesia (Active Comparator): General anesthesia
  Interventions: Drug: General anesthesia
- 2: Hypnosis (Experimental): Hypnosis with local anesthesia
  Interventions: Other: Local anesthetic + Hypnosis

INTERVENTIONS:
Other: Local anesthetic + Hypnosis — Modified state of consciousness allowing to be at the same time here and somewhere else. The individual is going to dive into his imagination to extract of an uncomfortable situation. And local anesthetic (solution of Xylocaine with adrenaline 1 % dabbed in 20 % of bicarbonate of sodium 4,2 %, maximal dose of 0,5ml / kg)
  Arms: 2: Hypnosis
Drug: General anesthesia — Sufentanil intravenous (0.1 in 0.2 µg / kg) and propofol (5 in 10 mg / kg on 3 mn) administration
  Arms: 1: General anesthesia

SUMMARY:
In adults, it is common to perform a number of superficial and non invasive surgeries under local anesthesia in order to limit the use of general anesthesia.

Hypnosis is a nonpharmacological therapies that can be used during surgery to improve the patient comfort and experience. The benefit of this practice has been widely demonstrated in adults, decreasing perioperative anxiety, postoperative pain scores as well as nausea and vomiting.

In pediatric surgery, hypnosis is an effective technique for the management of preoperative anxiety. It is used by many teams in their daily practice, particularly during anesthetic induction.

For 2 years, the team of pediatric anesthesia and surgery of the Montpellier University Hospital also offers for selected short and superficial non-invasive surgeries, an intraoperative management under hypnosis in association with ocal anesthesia as an alternative to general anesthesia. If this clinical practice of hypnosis is fully accepted and recognized in our intraoperative surgical unit, to date, no studies have evaluated the benefits of this technique compared to general anesthesia.

The objective of the study is to compare the impact of these techniques (hypnosis vs. general anesthesia) on postoperative experiences of children (rehabilitation time, anxiety, pain, nausea and vomiting, negative behavioral disorders).

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in infantile ambulatory surgery unit
* Patient whose general state corresponds to the classification of the American Society of Anesthesiologists (ASA) I to III
* Patient among whom the parents or the legal guardian gave their informed consent
* Patient member in a national insurance scheme

Exclusion Criteria:

* Patient presenting a contraindication to general anesthesia
* Patient presenting a contraindication to hypnosis (Chronic Encephalopathy with psychomotor delay, severe cognitive deficit, documented psychiatric disorders)

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-08-12 (Actual)

PRIMARY OUTCOMES:
Time to "home readiness" | up to 4 days
  The time to "home readiness" is defined when a patient is ready for discharge using an evidenced-based discharge scoring criteria.

SECONDARY OUTCOMES:
Postoperative pain | up to 10 minutes after the entrance to recovery room
  Pain is evaluated after surgery and each hour at hospital by the Faces Pain Scale - Revised (FPS-R).
Score Induction Compliance Checklist (ICC) | up to 10 minutes after the entrance to recovery room
Analgesic consumption | up to 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle CS Sola, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHRU Montpellier, Montpellier, France

REFERENCES:
- [Derived] Sola C, Devigne J, Bringuier S, Pico J, Coruble L, Capdevila X, Captier G, Dadure C. Hypnosis as an alternative to general anaesthesia for paediatric superficial surgery: a randomised controlled trial. Br J Anaesth. 2023 Mar;130(3):314-321. doi: 10.1016/j.bja.2022.11.023. Epub 2023 Jan 21. PMID 36690538